CLINICAL TRIAL: NCT04971330
Title: Evaluation of the Beckman Coulter Access Anti-HCV Assay as an Aid in the Diagnosis of HCV Infection: EU Clinical Trial Protocol
Brief Title: Access Anti-HCV Assay European Union (EU) Clinical Trial Protocol
Acronym: HCV-EU-10-18
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-TR18-0406
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: HCV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Known HCV Ab Positive Patients: leftover samples be tested with both reference anti-HCV assay and Access anti-HCV assay according to respective instructions for use (IFU) or study guide, as applicable, to determine non-reactive (NR), initial reactivity, and repeat reactivity. Reference assay will be Abbott Architect anti-HCV assay for positive samples.
  Interventions: Diagnostic Test: Access HCV
- Hospitalized Patients: leftover samples be tested with both reference anti-HCV assay and Access anti-HCV assay according to respective instructions for use (IFU) or study guide, as applicable, to determine non-reactive (NR), initial reactivity, and repeat reactivity. Reference assay will be Abbott Architect anti-HCV assay for hospitalized patient.
  For the specificity cohorts (blood donor and hospitalized patient samples), all HCV Ab positive results will have supplemental confirmation testing with HCV Immunoblot for final HCV Ab status
  Interventions: Diagnostic Test: Access HCV
- Unselected Blood Donors: Leftover samples be tested with both reference anti-HCV assay and Access anti-HCV assay according to respective instructions for use (IFU) or study guide, as applicable, to determine non-reactive (NR), initial reactivity, and repeat reactivity. les. For blood donors, Abbott PRISM HCV will be used as reference.
  For the specificity cohorts (blood donor and hospitalized patient samples), all HCV Ab positive results will have supplemental confirmation testing with HCV Immunoblot for final HCV Ab status.
  Interventions: Diagnostic Test: Access HCV

INTERVENTIONS:
Diagnostic Test: Access HCV — All samples were tested with both reference anti-HCV assay and Access anti-HCV assay according to respective instructions for use (IFU) or study guide, as applicable, to determine non-reactive (NR), initial reactivity, and repeat reactivity. Reference assay was Abbott Architect anti-HCV assay. For blood donors, Abbott PRISM HCV was used as reference.
  For the specificity cohorts (blood donor and hospitalized patient samples), all HCV Ab positive results will have supplemental confirmation testing with HCV Immunoblot for final HCV Ab status

SUMMARY:
The objective of this study was the collection and testing of clinical samples to determine the clinical performance in terms of diagnostic accuracy measured by specificity and sensitivity of the Access anti-Hepatitis C Virus (anti-HCV) assay on the DxI 9000 Access Immunoassay Analyzer. The Design Input Document (DID) indicates performance requirements and minimum target enrollment numbers (based on those in the CTS) of blood donor, hospitalized patient and known HCV antibody (Ab) positive samples for novel anti-HCV assays. A secondary objective was to determine the false initial reactive rate (IRR) of the Access anti-HCV assay.

DETAILED DESCRIPTION:
The study involved a multicenter, prospective and retrospective collection of samples, and testing of samples with the investigational Access anti-HCV assay. Subject sample enrollment was targeted to be approximately 8,000 specimens including approximately 6,000 blood donors and 1,500 hospitalized individuals for the specificity populations and 500 confirmed HCV Ab positive patients for the sensitivity population, required by European Union's Common Technical Specification for clinical validation of in vitro diagnostic medical devices and marketing needs to align with competitor submissions. Retrospective collection included HCV Ab positive genotyped samples from existing vendor collections meeting all inclusion/exclusion criteria.

All samples collected were anonymized, leftover, remnant samples and therefore member state or Institutional Review Board/Independent Ethics Committee approval was not required. Diagnostic sensitivity and specificity were evaluated for sample antibody status determined by a CE-marked anti-HCV assay (Abbott ARCHITECT anti-HCV assay for hospitalized patient and positive samples or Abbott PRISM HCV assay for blood donor samples) and Immunoblot testing with FUJIREBIO INNO-LIA HCV Score, if necessary. HCV RNA Polymerase Chain Reaction (PCR) or genotyping was requested or was available on all Immunoblot positive samples for further characterization, but these results were not used to determine final antibody status.

A portion of hospitalized patient samples (target 700/1500) and the majority of positive HCV Ab samples were collected and stored frozen prior to testing. A targeted portion of 800 hospitalized patient samples, 30 known positive samples and all blood donor samples were collected and tested fresh. Fresh blood donor and fresh hospitalized patient samples were used to determine false Initial Reactive Rate (IRR).

ELIGIBILITY:
Inclusion Criteria:

Anonymized or pseudo-anonymised leftover ethylenediaminetetraacetic acid (EDTA) plasma/serum samples from

* Males or females
* Aged ≥18 years of age
* Belonging to one of the following enrollment groups

  * Unselected blood donor
  * Hospitalized patient from GI, hepatology, Internal Medicine or Infectious Disease services
  * Known HCV Ab positive (by Immunoblot) at different stages of disease
* with at least 1.5 mL leftover sample (without genotype or PCR on same draw) OR
* at least 0.8 mL leftover sample (with genotype or HCV PCR on same draw)

Exclusion Criteria:

* Samples from subjects already included in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The test population includes :
  * 513 Known HCV Ab Positive Patients
  * 1533 Hospitalized patients
  * 5855 Unselected Blood donors
Sampling Method: Non-Probability Sample
Enrollment: 7901 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity | Baseline
  sensitivity and specificity relative to the final patient HCV Ab status determined from reference HCV Ab assay and/or supplemental confirmation testing (HCV Ab result by immunoblot).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Etablissement Français du Sang (EFS) Hauts-de-France - Normandie, Bois-Guillaume
  - Eurofins Biomnis, Ivry-sur-Seine
  - Cerba Xpert, Saint-Ouen-l'Aumône

IPD SHARING:
Plan to Share IPD: No